CLINICAL TRIAL: NCT01687361
Title: Can Branched Chain Amino Acids Supplementation Reduce Muscle Damage Induced by Neuromuscular Electrical Stimulation ? A Combined Functional and Metabolic Non-invasive Investigation in Healthy Humans.
Brief Title: Can Branched Chain Amino Acids Supplementation Reduce Muscle Damage Induced by Neuromuscular Electrical Stimulation? A Combined Functional and Metabolic Non-invasive Investigation in Healthy Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 2012-A00449-34; 2012-04 (Other: AP HM)
Record Dates: First submitted 2012-06-20; First posted 2012-09-18 (Estimated); Last update posted 2014-09-01 (Estimated); Status verified 2014-08

CONDITIONS: Neuromuscular Electrical Stimulation
MeSH Terms: interventions — Amino Acids, Branched-Chain; Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- branched-chain amino acids (BCAA) supplementation (Experimental)
  Interventions: Dietary Supplement: branched-chain amino acids (BCAA) supplementation
- PLACEBO (Placebo Comparator)
  Interventions: Drug: PLACEBO

INTERVENTIONS:
Dietary Supplement: branched-chain amino acids (BCAA) supplementation
  Arms: branched-chain amino acids (BCAA) supplementation
Drug: PLACEBO
  Arms: PLACEBO

SUMMARY:
Neuromuscular electrical stimulation (NMES) is commonly used in rehabilitation contexts in order to increase or restore muscle capacities of hypoactive patients or patients with articular trauma. Although this technique seems to be particularly adapted to muscle rehabilitation, growing evidence is emerging regarding potential damaging effects of electrically- induced isometric contractions in healthy humans. Recent studies have reported a 10 to 30-fold increase in creatine kinase (CK) activity coupled to significantly increased muscle soreness and impaired force production as a result of NMESs. On that basis, further studies should be conducted on these deleterious effects which might limit the clinical application of NMES.

Over the last decade, many studies paid attention to branched-chain amino acids (BCAA) supplementation as a potential prophylactic/therapeutic approach. The rationale of this approach is that BCAA might increase protein synthesis and reduce protein breakdown through physiological mechanisms involving mTOR regulation pathway (mammalian Target of Rapamycin). Additionally, BCAA could also be used as energetic substrate during exercise when glycogen stores are depleted. Overall, previous results have supported the efficacy of BCAA supplementation in attenuating muscle damage. Nevertheless, comprehensive studies investigating the effect of amino acid supplementation on markers of muscle damage are still scarce.

Magnetic resonance imaging (IRM) and phosphorus 31 magnetic resonance spectroscopy (31P-MRS) are powerful non invasive tools allowing the exploration of skeletal muscle structure and energy metabolism.

This ambitious project is devoted to the anatomical, functional and metabolic characterization of BCAA supplementation after NMES using MRI and 31P-MRS. Various markers of muscle damage, including maximal voluntary force production, T2 values and apparent diffusion coefficient (obtained by MRI) and energy metabolism assessed at rest and during exercise (using 31P-MRS), will be obtained before and after NMES. This project is of utmost importance for improving our knowledge of anatomic, metabolic and functional events related to BCAA supplementation in the context of exercise-induced muscle damage

ELIGIBILITY:
Inclusion Criteria:

* Male
* Between 18 and 35 years
* Subjects will have to be unhurt:

  * Any general disease
  * Psychiatric disorders(confusions)
  * Any infectious, inflammatory, tumoral, vascular, degenerative or traumatic pathology
* They will have to follow no chronic treatment
* They will have to be unhurt of any history of alcoholism or drug addiction

Exclusion Criteria:

* Contraindications for an examination MRI
* Suffering from claustrophobia
* Having stimulating one cardiac, carriers of a system Holter, carriers of hook(staple) (clip) surgical metallic, carriers of a prosthesis or a metallic implant (or quite other metallic foreign bodies), carriers of a prosthesis dental (device), carriers of a hearing aid, carriers of an insulin pump
* Having been hurt by pieces of shrapnel or lead
* Having had a dislocation, a fracture or a recent surgical operation (less than 6 months before the inclusion)
* Having followed a treatment with anti-inflammatory drugs during the last 3 months
* Having followed a treatment with amino acids during the last 3 months
* Having followed a treatment(processing) with anabolic steroids during the last 3 months
* Having participated in a program of body-building of lower limbs during the last 6 months

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2012-06; Primary Completion 2013-06 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
evaluation of the muscular responsiveness | 24 MONTHS

SECONDARY OUTCOMES:
evaluation of the effects of a supplementation in AAB | 24 MONTTHS
  on the physiological aspects

CONTACTS AND LOCATIONS:
Overall Officials: BERNARD BELAIGUES, Study Director — Assistance Publique hôpitaux de Marseille; jean pierre mattei, Principal Investigator — AP HM
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France